CLINICAL TRIAL: NCT07269470
Title: Phase II Study Assessing the Safety and Efficacy of Dasatinib in Combination With Ropeginterferon in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1526; NCI-2025-08780 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 2 Treatment with Dasatinib (PO) + Ropeginterferon (SC) (Experimental): Participants will receive treatment on an outpatient basis.
  Interventions: Drug: Dasatinib; Drug: Ropeginterferon alfa-2b (P1101)

INTERVENTIONS:
Drug: Dasatinib — Given orally daily for 3 cycles
  Other Names: Sprycel
Drug: Ropeginterferon alfa-2b (P1101) — Given subcutaneous through injection

SUMMARY:
The goal of this clinical research study is to find out if treatment with a combination of dasatinib plus ropeginterferon can help to control CML-CP. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

To assess the rate of molecular response 4.5 (4.5 log-reduction of BCR::ABL1 transcripts or level ≤ 0.0032% IS) by 12 months of therapy

Secondary Objectives:

To assess the rate of complete cytogenetic response (BCR::ABL1 transcripts ≤ 1% IS) by 12 months of therapy

To assess the rate of major molecular response (BCR::ABL1 transcripts ≤ 0.1% IS) by 12 months of therapy

To estimate the proportion of patients achieving MR4.5 at 6, 18, 24, and 36 months of therapy

To estimate the rate of sustained deep molecular response (DMR; BCR::ABL1 transcripts ≤ 0.01% IS) for 2 years and longer

To evaluate the safety of the combination

To assess event-free survival and overall survival for 10 years after the last patient is enrolled

ELIGIBILITY:
Inclusion Criteria:

Adult patients age ≥18 years.

Patients must have a diagnosis of Ph-positive or BCR::ABL1 positive CML in chronic phase.

Patients who received prior hydroxyurea, 1 to 2 doses of cytarabine, and/or an FDA approved TKI for <30 days are eligible.

Patients with additional chromosomal abnormalities at diagnosis (early disease) and no other criteria for accelerated phase will be eligible for this study.

ECOG performance status ≤2.

Patients must have adequate end organ function, defined as the following: total bilirubin

≤1.5x ULN (unless secondary to Gilbert's disease, in which case should be ≤2.5x ULN), SGPT or SGOT ≤3x ULN, creatinine clearance ≥30mL/min calculated using modified Cockcroft-Gault.

Ability to understand and the willingness to sign a written informed consent document.

Dasatinib is known to be teratogenic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better.

Exclusion Criteria:

Patients who have received more than 30 days of prior FDA approved TKI or more than 2 doses of cytarabine.

Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.

Patients who are receiving any other investigational agents.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib, ropeginterferon, or other agents used in study.

NYHA cardiac class III-IV heart disease.

Active autoimmune disease at screening.

History or presence of clinically relevant depression

Patients with active, uncontrolled psychiatric disorders including psychosis, major depression, and bipolar disorders.

Patients with cognitive impairment or psychiatric illness/social situations that would limit compliance with study requirements.

Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment and having detectable virus load. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface antigen negative, anti-HBs antibody positive and antihepatitis B core antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins may participate.

Any contraindications or hypersensitivity to dasatinib or IFN-α and/or its excipients

Patients in accelerated (except as noted in inclusion criteria 4.1) or blast phase are excluded.

Pregnant women are excluded from this study because dasatinib is an agent with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Haddad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org